CLINICAL TRIAL: NCT02388945
Title: Validity and Security of Domestic Automated Peritoneal Dialysis Machine: A Prospective, Randomized, Controlled, Multi-Center Clinical Trial
Brief Title: A Study of Domestic Automated Peritoneal Dialysis Machine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Usix-APD-001
Record Dates: First submitted 2015-02-15; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Disorders Associated With Peritoneal Dialysis
MeSH Terms: interventions — Peritoneal Dialysis, Continuous Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A APDGroup (Experimental): PDGO APD machines used in the PD patients for 8 weeks
  Interventions: Other: APD
- B CAPDGroup (Active Comparator): CAPD used in the PD Patients for 8 weeks
  Interventions: Other: CAPD

INTERVENTIONS:
Other: APD — PDGO APD machines used in the PD patients for 8 weeks
  Arms: A APDGroup
Other: CAPD — CAPD used in the PD Patients for 8 weeks
  Arms: B CAPDGroup

SUMMARY:
This prospective, randomized, controlled, multi-center clinical trial will evaluate the validity and security of domestic APD machine compared with the patients followed CAPD.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) is one of important way of renal replacement treatment worldwide. In China, about 40,000 patients suffered from end stage renal disease treated with PD, and almost of them followed continuous ambulatory peritoneal dialysis (CAPD) because of the expensive price of import automated PD (APD) machines although the higher clearance of solute, lower rate of PD related peritonitis and higher quality of life (QOL) in patients treated with APD compared those with CAPD. Now, cheaper domestic APD machines ( PDGO, Fuzhou, China) are accessed to the ESRD patients in china, but the efficacy and safety of which are not fully clear. This will be a prospective, randomized, controlled, multi-center study. Patients in treatment group will receive APD while those in control group will receive CAPD for 8 weeks. After followed-up for 8 weeks, the adequacy of PD, residual kidney function , peritoneum function and QOL of patients will be evaluated.

ELIGIBILITY:
Inclusion criteria:

1. The duration of PD is more than 1 month.
2. The age is range from 18 to 80 years old.
3. The patient can be treated with regular PD in home.
4. The volume of peritoneal dialysate is from 8L to 10 L in 1 day.
5. The patient can be visited regularly.
6. The patient must be freely given informed consent

Exclusion criteria:

1. Peritonitis was happened within 1 month
2. The KT/V<1.7
3. Infections in the exit or tunnel
4. With tumors.
5. With low transport of peritoneum.
6. With mental and behavior disorders.
7. With acute renal failure
8. Hemodialysis meanwhile
9. With heart failure( NYHA III-IV ) or cardio- cerebrovascular events
10. Attending other clinical trails
11. Refused to give informed consent Exit criteria

（1）Stop PD for more than 10 days （2）The patient demand to quit from the RCT （3）With serious adverse events.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Adequacy of dialysis | up to 8 weeks
  kt/v

SECONDARY OUTCOMES:
Residual kidney function | up to 6 months
  Residual kidney kt/v
Peritoneal function | up to 6 months
  Peritoneal equilibration test

CONTACTS AND LOCATIONS:
Overall Officials: Zongpei Jiang, M.D. & Ph.D., Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of Nephrology, 6th Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China